CLINICAL TRIAL: NCT05315583
Title: Study of the Neutralizing Power of Anti-SARS-CoV-2 (Anti-COVID-19) Serum Antibodies
Brief Title: Neutralizing Power of Anti-SARS-CoV-2 (Anti-COVID-19) Serum Antibodies
Acronym: PNAS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Now that the COVID period has passed, patient recruitment has fallen off.
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHRO-2022-03
Record Dates: First submitted 2022-03-16; First posted 2022-04-07 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: COVID-19; SARS CoV 2 Infection
Keywords: COVID-19; Vaccines; Monoclonal antibodies; Neutralization; Serum; Nasal mucosa
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Collection of biological samples (Day 0, D3, D15, Month 1, M2, M3, M4, M5, M6, M9, M12, M18) with associated data for the study of the kinetics of antibodies against COVID-19. All participants will have at each of the visits: a venipuncture sample of 2 dry tubes of 7 mL to make up 3 aliquots and a nasopharyngeal swab (optional). The aliquots of serum / plasma and the nasopharyngeal swab will be stored at -80°C until sent to the Pasteur Institute.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group with collection of biological samples (Other): All participants will have at each of the visits: a venipuncture sample of 2 dry tubes of 7 mL to make up 3 aliquots and a nasopharyngeal swab (optional). The aliquots of serum / plasma and the nasopharyngeal swab will be stored at -80°C until sent to the Pasteur Institute.
  Interventions: Other: Collection of biological samples

INTERVENTIONS:
Other: Collection of biological samples — All participants will have at each of the visits: a venipuncture sample of 2 dry tubes of 7 mL to make up 3 aliquots and a nasopharyngeal swab (optional). The aliquots of serum / plasma and the nasopharyngeal swab will be stored at -80°C until sent to the Pasteur Institute.

SUMMARY:
Natural infection, vaccines and treatments (like monoclonal antibodies) lead to the appearance of a neutralizing power in the serum (due to induced or injected antibodies). This neutralizing power is recognized as a correlate of protection against a (new) infection. This study aims to measure the neutralizing power of the serum of patients (whether or not they have been infected with SARS-CoV-2) according to the treatments and/or vaccines received and to assess the durability of this power in the time.

DETAILED DESCRIPTION:
Infection, vaccines and treatments (like monoclonal antibodies) lead to the appearance of a neutralizing power in the serum (due to induced or injected antibodies). This neutralizing power is recognized as a correlate of protection against (new) infection. The purpose of this study is to measure the neutralizing power of the serum of patients (whether or not they have been infected with SARS-CoV-2) depending on the treatments and/or vaccines received and to assess the durability of this power over time.

The main objective is to measure and describe the evolution of the serum humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies (vaccines - whatever the mode of action -, monoclonal antibodies).

The secondary objectives are:

* to measure and describe the antibody response at the level of the nasal mucosa (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies, collected by means of a nasal swab) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies SARS-CoV-2.
* to describe the incidence of COVID in the study patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult volunteers for the study, having received or about to receive any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies (vaccines - whatever the mode of action -, monoclonal antibodies).
* Having given their consent to participate in the study

Exclusion Criteria:

* Minors
* Pregnant women
* Persons under tutorship or curatorship
* Protected adults
* Person under legal protection
* Person not affiliated to a social security scheme
* Persons unable to express their consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2023-03-16 (Actual)

PRIMARY OUTCOMES:
Evolution of the serum humoral response | Day 0
  Evolution of the serum humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Flow in BAU/ml (Binding Antibody Unit/milliliter)
Evolution of the serum humoral response | Day 0
  Evolution of the serum humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Fuse in ED50 (Effective Dilution 50% titers)
Evolution of the serum humoral response | Day 3
  Evolution of the serum humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Flow in BAU/ml (Binding Antibody Unit/milliliter)
Evolution of the serum humoral response | Day 3
  Evolution of the serum humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Fuse in ED50 (Effective Dilution 50% titers)
Evolution of the serum humoral response | Day 15
  Evolution of the serum humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Flow in BAU/ml (Binding Antibody Unit/milliliter)
Evolution of the serum humoral response | Day 15
  Evolution of the serum humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Fuse in ED50 (Effective Dilution 50% titers)
Evolution of the serum humoral response | Month 1
  Evolution of the serum humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Flow in BAU/ml (Binding Antibody Unit/milliliter)
Evolution of the serum humoral response | Month 1
  Evolution of the serum humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Fuse in ED50 (Effective Dilution 50% titers)
Evolution of the serum humoral response | Month 2
  Evolution of the serum humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Flow in BAU/ml (Binding Antibody Unit/milliliter)
Evolution of the serum humoral response | Month 2
  Evolution of the serum humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Fuse in ED50 (Effective Dilution 50% titers)
Evolution of the serum humoral response | Month 3
  Evolution of the serum humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Flow in BAU/ml (Binding Antibody Unit/milliliter)
Evolution of the serum humoral response | Month 3
  Evolution of the serum humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Fuse in ED50 (Effective Dilution 50% titers)
Evolution of the serum humoral response | Month 4
  Evolution of the serum humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Flow in BAU/ml (Binding Antibody Unit/milliliter)
Evolution of the serum humoral response | Month 4
  Evolution of the serum humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Fuse in ED50 (Effective Dilution 50% titers)
Evolution of the serum humoral response | Month 5
  Evolution of the serum humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Flow in BAU/ml (Binding Antibody Unit/milliliter)
Evolution of the serum humoral response | Month 5
  Evolution of the serum humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Fuse in ED50 (Effective Dilution 50% titers)
Evolution of the serum humoral response | Month 6
  Evolution of the serum humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Flow in BAU/ml (Binding Antibody Unit/milliliter)
Evolution of the serum humoral response | Month 6
  Evolution of the serum humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Fuse in ED50 (Effective Dilution 50% titers)
Evolution of the serum humoral response | Month 9
  Evolution of the serum humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Flow in BAU/ml (Binding Antibody Unit/milliliter)
Evolution of the serum humoral response | Month 9
  Evolution of the serum humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Fuse in ED50 (Effective Dilution 50% titers)
Evolution of the serum humoral response | Month 12
  Evolution of the serum humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Flow in BAU/ml (Binding Antibody Unit/milliliter)
Evolution of the serum humoral response | Month 12
  Evolution of the serum humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Fuse in ED50 (Effective Dilution 50% titers)
Evolution of the serum humoral response | Month 18
  Evolution of the serum humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Flow in BAU/ml (Binding Antibody Unit/milliliter)
Evolution of the serum humoral response | Month 18
  Evolution of the serum humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Fuse in ED50 (Effective Dilution 50% titers)

SECONDARY OUTCOMES:
Evolution of the mucosal humoral response | Day 0
  Evolution of the mucosal humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Flow in BAU/ml (Binding Antibody Unit/milliliter)
Evolution of the mucosal humoral response | Day 0
  Evolution of the mucosal humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Fuse in ED50 (Effective Dilution 50% titers)
Evolution of the mucosal humoral response | Day 3
  Evolution of the mucosal humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Flow in BAU/ml (Binding Antibody Unit/milliliter)
Evolution of the mucosal humoral response | Day 3
  Evolution of the mucosal humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Fuse in ED50 (Effective Dilution 50% titers)
Evolution of the mucosal humoral response | Day 15
  Evolution of the mucosal humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Flow in BAU/ml (Binding Antibody Unit/milliliter)
Evolution of the mucosal humoral response | Day 15
  Evolution of the mucosal humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Fuse in ED50 (Effective Dilution 50% titers)
Evolution of the mucosal humoral response | Month 1
  Evolution of the mucosal humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Flow in BAU/ml (Binding Antibody Unit/milliliter)
Evolution of the mucosal humoral response | Month 1
  Evolution of the mucosal humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Fuse in ED50 (Effective Dilution 50% titers)
Evolution of the mucosal humoral response | Month 2
  Evolution of the mucosal humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Flow in BAU/ml (Binding Antibody Unit/milliliter)
Evolution of the mucosal humoral response | Month 2
  Evolution of the mucosal humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Fuse in ED50 (Effective Dilution 50% titers)
Evolution of the mucosal humoral response | Month 3
  Evolution of the mucosal humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Flow in BAU/ml (Binding Antibody Unit/milliliter)
Evolution of the mucosal humoral response | Month 3
  Evolution of the mucosal humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Fuse in ED50 (Effective Dilution 50% titers)
Evolution of the mucosal humoral response | Month 4
  Evolution of the mucosal humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Flow in BAU/ml (Binding Antibody Unit/milliliter)
Evolution of the mucosal humoral response | Month 4
  Evolution of the mucosal humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Fuse in ED50 (Effective Dilution 50% titers)
Evolution of the mucosal humoral response | Month 5
  Evolution of the mucosal humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Flow in BAU/ml (Binding Antibody Unit/milliliter)
Evolution of the mucosal humoral response | Month 5
  Evolution of the mucosal humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Fuse in ED50 (Effective Dilution 50% titers)
Evolution of the mucosal humoral response | Month 6
  Evolution of the mucosal humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Flow in BAU/ml (Binding Antibody Unit/milliliter)
Evolution of the mucosal humoral response | Month 6
  Evolution of the mucosal humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Fuse in ED50 (Effective Dilution 50% titers)
Evolution of the mucosal humoral response | Month 9
  Evolution of the mucosal humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Flow in BAU/ml (Binding Antibody Unit/milliliter)
Evolution of the mucosal humoral response | Month 9
  Evolution of the mucosal humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Fuse in ED50 (Effective Dilution 50% titers)
Evolution of the mucosal humoral response | Month 12
  Evolution of the mucosal humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Flow in BAU/ml (Binding Antibody Unit/milliliter)
Evolution of the mucosal humoral response | Month 12
  Evolution of the mucosal humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Fuse in ED50 (Effective Dilution 50% titers)
Evolution of the mucosal humoral response | Month 18
  Evolution of the mucosal humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Flow in BAU/ml (Binding Antibody Unit/milliliter)
Evolution of the mucosal humoral response | Month 18
  Evolution of the mucosal humoral response (titer and neutralizing capacity of anti-SARS-CoV-2 antibodies) following any intervention inducing or conferring neutralizing anti-SARS-CoV-2 antibodies.
  S-Fuse in ED50 (Effective Dilution 50% titers)
Proportion of participants developing COVID-19 infection after these treatments | Day 0
  Proportion of participants developing COVID-19 infection after these treatments documented (by specific PCR) SARS-CoV-2 infection.
Proportion of participants developing COVID-19 infection after these treatments | Day 3
  Proportion of participants developing COVID-19 infection after these treatments documented (by specific PCR) SARS-CoV-2 infection.
Proportion of participants developing COVID-19 infection after these treatments | Day 15
  Proportion of participants developing COVID-19 infection after these treatments documented (by specific PCR) SARS-CoV-2 infection.
Proportion of participants developing COVID-19 infection after these treatments | Month 1
  Proportion of participants developing COVID-19 infection after these treatments documented (by specific PCR) SARS-CoV-2 infection.
Proportion of participants developing COVID-19 infection after these treatments | Month 2
  Proportion of participants developing COVID-19 infection after these treatments documented (by specific PCR) SARS-CoV-2 infection.
Proportion of participants developing COVID-19 infection after these treatments | Month 3
  Proportion of participants developing COVID-19 infection after these treatments documented (by specific PCR) SARS-CoV-2 infection.
Proportion of participants developing COVID-19 infection after these treatments | Month 4
  Proportion of participants developing COVID-19 infection after these treatments documented (by specific PCR) SARS-CoV-2 infection.
Proportion of participants developing COVID-19 infection after these treatments | Month 5
  Proportion of participants developing COVID-19 infection after these treatments documented (by specific PCR) SARS-CoV-2 infection.
Proportion of participants developing COVID-19 infection after these treatments | Month 6
  Proportion of participants developing COVID-19 infection after these treatments documented (by specific PCR) SARS-CoV-2 infection.
Proportion of participants developing COVID-19 infection after these treatments | Month 9
  Proportion of participants developing COVID-19 infection after these treatments documented (by specific PCR) SARS-CoV-2 infection.
Proportion of participants developing COVID-19 infection after these treatments | Month 12
  Proportion of participants developing COVID-19 infection after these treatments documented (by specific PCR) SARS-CoV-2 infection.
Proportion of participants developing COVID-19 infection after these treatments | Month 18
  Proportion of participants developing COVID-19 infection after these treatments documented (by specific PCR) SARS-CoV-2 infection.

CONTACTS AND LOCATIONS:
Overall Officials: Thierry PRAZUCK, Dr, Principal Investigator — CHR d'Orléans
Locations (1):
- Centre Hospitalier Régional d'Orléans, France, Orléans, France

REFERENCES:
- [Background] Grzelak L, Temmam S, Planchais C, Demeret C, Tondeur L, Huon C, Guivel-Benhassine F, Staropoli I, Chazal M, Dufloo J, Planas D, Buchrieser J, Rajah MM, Robinot R, Porrot F, Albert M, Chen KY, Crescenzo-Chaigne B, Donati F, Anna F, Souque P, Gransagne M, Bellalou J, Nowakowski M, Backovic M, Bouadma L, Le Fevre L, Le Hingrat Q, Descamps D, Pourbaix A, Laouenan C, Ghosn J, Yazdanpanah Y, Besombes C, Jolly N, Pellerin-Fernandes S, Cheny O, Ungeheuer MN, Mellon G, Morel P, Rolland S, Rey FA, Behillil S, Enouf V, Lemaitre A, Creach MA, Petres S, Escriou N, Charneau P, Fontanet A, Hoen B, Bruel T, Eloit M, Mouquet H, Schwartz O, van der Werf S. A comparison of four serological assays for detecting anti-SARS-CoV-2 antibodies in human serum samples from different populations. Sci Transl Med. 2020 Sep 2;12(559):eabc3103. doi: 10.1126/scitranslmed.abc3103. Epub 2020 Aug 17. PMID 32817357
- [Background] Planas D, Bruel T, Grzelak L, Guivel-Benhassine F, Staropoli I, Porrot F, Planchais C, Buchrieser J, Rajah MM, Bishop E, Albert M, Donati F, Prot M, Behillil S, Enouf V, Maquart M, Smati-Lafarge M, Varon E, Schortgen F, Yahyaoui L, Gonzalez M, De Seze J, Pere H, Veyer D, Seve A, Simon-Loriere E, Fafi-Kremer S, Stefic K, Mouquet H, Hocqueloux L, van der Werf S, Prazuck T, Schwartz O. Sensitivity of infectious SARS-CoV-2 B.1.1.7 and B.1.351 variants to neutralizing antibodies. Nat Med. 2021 May;27(5):917-924. doi: 10.1038/s41591-021-01318-5. Epub 2021 Mar 26. PMID 33772244
- [Derived] Clairon Q, Prague M, Planas D, Bruel T, Hocqueloux L, Prazuck T, Schwartz O, Thiebaut R, Guedj J. Modeling the kinetics of the neutralizing antibody response against SARS-CoV-2 variants after several administrations of Bnt162b2. PLoS Comput Biol. 2023 Aug 7;19(8):e1011282. doi: 10.1371/journal.pcbi.1011282. eCollection 2023 Aug. PMID 37549192